CLINICAL TRIAL: NCT03771131
Title: A Group Study on the Effects of a Short Multi-Domain Cognitive Training in Healthy Elderly Italian People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Roberta Daini, Professor, University of Milano Bicocca
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DD
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Age-related Cognitive Decline
Keywords: healthy cognitive ageing; multi-domain cognitive training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Group receiving the multi-domain cognitive training
  Interventions: Behavioral: Multi-domain cognitive training
- Control group (No Intervention): Passive control group

INTERVENTIONS:
Behavioral: Multi-domain cognitive training — Weekly sessions of multi-domain cognitive training, each lasting around one hour for an overall duration of the training of 3 months (13 sessions)
  Arms: Experimental group

SUMMARY:
Alongside physiological cognitive ageing, nowadays there is an alarming increase in the incidence of dementia that requires communities to invest in its prevention. The engagement in cognitively stimulating activities and strong social networks have been identified among those protective factors promoting successful cognitive ageing. One aspect regarding cognitive stimulation concerns the relevance of the frequency of an external intervention. For these reasons, the aim of this study was to evaluate the efficacy of a 3-month multi-domain cognitive training program, administered once per week in a group of healthy elderly aged over 60 years old. Their results obtained on a series of neuropsychological tests, both pre- (t0) and post-training (t1), were compared with those of a passive control group who did not receive the cognitive training.

DETAILED DESCRIPTION:
Participants were assigned to the experimental or control group based on their time of application to the program. Both experimental and control group underwent a neuropsychological assessment to investigate different cognitive domains, before and after (~3 months) the training program. Based on the scores obtained during the preliminary neuropsychological assessment, the participants of the experimental training group were divided into small subgroups (ranging from 8 to 12 subjects) to further address individualization of training (i.e. level of difficulty of the exercises proposed). The experimental group attended weekly sessions of the multi-domain cognitive training. Each session lasted around one hour and the overall duration of the training was of 3 months, for a total of 13 sessions. To promote improvement transfer to everyday life, some of the exercises proposed were ecological in their nature, in that, they asked participants to solve tasks that recalled everyday situations (such as remembering names or road maps). Furthermore, throughout the training, approximately once every two sessions brief psycho-educational interventions were provided.

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years

Exclusion Criteria:

* Negative anamnesis for neurological and/or psychiatric diseases
* No suspected cognitive impairment as assessed during the pre-training neuropsychological testing (>2 pathological scores)

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
Mean change from pre-training in Montreal Congnitive Assessment (MoCA) scores | Pre- and post-training (after ~3 months of training)
  Raw score, assessing global cognitive functioning. Cutoff: < 17.362. Cutoff scores indicate the value above/below which the cognitive performance is considered pathological.
Mean change from pre-training in Forward and Backward Digit and Corsi Span scores | Pre- and post-training (after ~3 months of training)
  Raw score, assessing verbal and visuo-spatial short term memory. Cutoff: < 4.26 (Forward Digit Span), < 2.65 (Backward Digit Span), < 3.46 (Forward Corsi Span), < 3.08 (Backward Corsi Span). Cutoff scores indicate the value above/below which the cognitive performance is considered pathological.
Mean change from pre-training in Short Story test scores | Pre- and post-training (after ~3 months of training)
  Raw score, assessing verbal long term memory. Cutoff: < 7.5. Cutoff scores indicate the value above/below which the cognitive performance is considered pathological.
Mean change from pre-training in Copy and Recall of Rey-Osterrieth Complex Figure scores | Pre- and post-training (after ~3 months of training)
  Raw score, assessing constructional abilities and visuo-spatial long term memory. Cutoff: < 28.87 (Copy), < 9.46 (Recall). Cutoff scores indicate the value above/below which the cognitive performance is considered pathological.
Mean change from pre-training in Semantic and Phonological Verbal Fluency scores | Pre- and post-training (after ~3 months of training)
  Raw score, assessing executive functions. Cutoff: < 16 (Phonological), < 24 (Semantic). Cutoff scores indicate the value above/below which the cognitive performance is considered pathological.
Mean change from pre-training in Stroop color and word test scores | Pre- and post-training (after ~3 months of training)
  Raw score, assessing inhibitory control. Cutoff: > 36.92 (for Time measure), > 4.24 (for Error measure). Cutoff scores indicate the value above/below which the cognitive performance is considered pathological.
Mean change from pre-training in Trail Making test scores | Pre- and post-training (after ~3 months of training)
  Raw score, assessing attention. Cutoff: > 93 (TMT A), > 282 (TMT B), > 186 (TMT B-A). Cutoff scores indicate the value above/below which the cognitive performance is considered pathological.
Mean change from pre-training in Raven's coloured matrices scores | Pre- and post-training (after ~3 months of training)
  Raw score, assessing non-verbal reasoning. Cutoff: < 18. Cutoff scores indicate the value above/below which the cognitive performance is considered pathological.

SECONDARY OUTCOMES:
Mean scores in the Post-training questionnaire | Post-training (after ~3 months of training)
  Scores assessing both the satisfaction level about the training and the possible impact of the program on participants' everyday activities, mood and socialization. Each question was measured on a 5-point Likert scale (1: most negative score; 5: most positive score).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Milan-Bicocca, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tagliabue CF, Guzzetti S, Gualco G, Boccolieri G, Boccolieri A, Smith S, Daini R. A group study on the effects of a short multi-domain cognitive training in healthy elderly Italian people. BMC Geriatr. 2018 Dec 27;18(1):321. doi: 10.1186/s12877-018-1014-x. PMID 30587151